CLINICAL TRIAL: NCT01120067
Title: Intensive Treatment of Chronic Pain and PTSD for OEF/OIF Veterans
Brief Title: Intensive Treatment for Chronic Pain and Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6281-I
Record Dates: First submitted 2010-04-30; First posted 2010-05-10 (Estimated); Results first posted 2016-12-16 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Psychology; Pain; Veterans; Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Treatment (Experimental): Intensive 3 week treatment for pain and PTSD. This includes elements of Cognitive Processing Therapy and CBT for Chronic Pain
  Interventions: Behavioral: Intensive Treatment
- Treatment as Usual (Experimental): Treatment as Usual. Participants are eligible for all treatment services as needed except for treatment of pain or PTSD
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Intensive Treatment — Participants randomized to the Intensive Treatment condition will attend 6 bi-weekly outpatient therapy sessions conducted in an individual format of 90 minutes in duration.
  Arms: Intensive Treatment
Behavioral: Treatment as Usual — Treatment as Usual.
  Arms: Treatment as Usual

SUMMARY:
This study is investigating the efficacy of an intensive (3 week) integrated treatment for Veterans with both pain and PTSD.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to evaluate the efficacy of an intensive integrated treatment for Veterans with comorbid chronic pain and posttraumatic stress disorder (PTSD). A secondary objective is to examine potential mechanisms of action that might account for improvements in pain or PTSD. Third, exploratory analyses will be conducted to assess the relationship between participation in treatment and cognitive functioning. It is hypothesized that 1) participants receiving the intensive treatment (PT) will report significantly greater decreases in symptoms of pain and PTSD from pre-treatment to post-treatment when compared to participants randomized to a standard care (SC) condition, and 2) participants receiving PT will show greater maintenance of change on measures of pain and PTSD at 3 months following the completion of treatment when compared to participants randomized to the SC condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible to participate if they have constant pain of at least three months duration with a neurologic or musculoskeletal etiology.
* Patients must also meet diagnostic criteria for PTSD.

Exclusion Criteria:

* Patients with life threatening or acute physical illness, current alcohol or substance abuse, current psychosis or suicidal ideation, and individuals seeking pain treatment such as surgical interventions will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-08-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2016-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Otis, BS BA PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsai J, Whealin JM, Scott JC, Harpaz-Rotem I, Pietrzak RH. Examining the relation between combat-related concussion, a novel 5-factor model of posttraumatic stress symptoms, and health-related quality of life in Iraq and Afghanistan veterans. J Clin Psychiatry. 2012 Aug;73(8):1110-8. doi: 10.4088/JCP.11m07587. Epub 2012 Jun 26. PMID 22781019

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Treatment | Treatment as Usual
Started | 12 | 11
Completed | 7 | 10
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — fail to engage >3 sessions | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intensive Treatment | Treatment as Usual | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.75 (10.39) | 52.09 (10.64) | 49.79 (10.274)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 12 | 9 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 9 | 9 | 18
  African American | 2 | 2 | 4
  Hispanic | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 11 | 23

OUTCOME MEASURES:

1. Primary Outcome: McGill Pain Questionnaire
Description: McGill Pain Questionnaire (MPQ; Melzack, 1975): is a self-report questionnaire consisting of 102 words separated into three major classes; the sensory, affective, and evaluative aspects of pain. Respondents are asked to circle the word that best describes their pain. The stability, reliability, and validity of the MPQ have been established (Reading, Everitt, & Sledmere, 1982). The MPQ total score ranges from 0 to 78 with higher values indicating more significant pain.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intensive Treatment | Treatment as Usual
Number analyzed (Participants) | 12 | 11
units on a scale | 31.91 (13.55) | 30.83 (13.61)

ADVERSE EVENTS:
Arm/Group | Intensive Treatment | Treatment as Usual
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

LIMITATIONS AND CAVEATS:
Small N due to challenges associated with recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No